CLINICAL TRIAL: NCT03970135
Title: Fedt og Sukkerstofskiftet Under Faste Hos Patienter Med Lav Muskelmasse.
Brief Title: Fat and Glucose Metabolism in Fed and Fasted State in Patients With Low Skeletal Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mette Cathrine Oerngreen, PI, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-16049377
Record Dates: First submitted 2019-05-21; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Spinal Muscular Atrophy; Merosin Deficient Congenital Muscular Dystrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular dystrophy congenital, merosin negative | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Experimental)
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Fasting for 24 hours or until hypoglycemia (blood glucose < 3mmol/L) or symptoms of hypoglycemia

SUMMARY:
In a study from 2003 the investigators showed that adult patients with very low skeletal muscle mass (spinal muscular atrophy (SMA) type II, Duchenne muscular dystrophy, congenital muscular dystrophy) are prone to develop hypoglycemia during prolonged fasting. Since then case reports have described the same phenomenon with hypoglycemia and metabolic crises in children with low skeletal muscle mass provoked by infection, fasting and surgery. Pathophysiological mechanisms of metabolism have never been investigated in adults or children with SMA II. Thus the investigators studied fat and glucose metabolism during prolonged fasting in patients with SMA II and LAMA 2 and compared results to those found in healthy controls.

DETAILED DESCRIPTION:
Design. This is a prospective case-control study investigating fat and glucose metabolism in patients with low muscle mass during prolonged fasting, comparing results to those found in healthy controls.

Setting. All children were admitted to the Department of Pediatrics and Adolescents medicine, Rigshospitalet, and all adult subjects were admitted to the Department of Neurology, Rigshospitalet at 4 pm for a 24-hour fasting period.

Protocol. The protocol consisted of two visits. A pre-experimental visit and a study visit.

Pre-experimental visit. Total muscle mass presented as lean body mass (LBM) was measured by DEXA scan. Furthermore, pre-experimental preparations included that all subjects were instructed to follow national nutritional recommendations with a healthy diet consisting of less than 30% fat, low fat protein, long chain carbohydrates and minimize sugar intake three days before the study.

Study visit. Patients were admitted to the hospital at 16:00 hours for IV catheter placement and a standardized evening meal at 17:00. Two venous catheters were inserted, one in the cubital vein (for stable-isotope infusion) and one in the distal cephalic vein (for blood sampling). A heating pad, covering the hand and distal forearm, ensured shunting of arterial blood to the veins in order to obtain arterialized blood. A primed, constant rate infusion of [U-13C]-palmitate (0.0026 mg kg-1 min-1, primed by a 0.085 mg kg-1 NaH13CO3 bolus) and [D2]-glucose (0.0728 mg kg-1 min-1, primed by a 3.203 mg kg-1 D2- glucose bolus) was delivered by a Gemini PC2 pump (IMED, San Diego, CA). Preparation of tracers and tracer calculations were performed as described.

Blood and air samples were collected just before start of infusion of the stable isotopes, and again after 2, 10, 14, 16, 18, 20, 22 and 24 hours of fasting (figure 1). Gas exchange measurements (indirect calorimetry) were performed with a metabolic cart (Cosmed Quark b2; Cosmed Srl., Milan, Italy). At the same time-points, expired air was collected in a 15 L Douglas bag (Hans Rudolph, Kansas City, MO, USA) and 10 mL samples were transferred to vacuum tubes (Vacutainer, BD, Franklin Lakes, NJ, USA) for 13CO2 analysis.

The blood glucose levels were monitored continuously at all blood sampling times and every third hour during the night in the patients. If the subjects developed symptoms of hypoglycaemia (fatigue, dizziness, nausea) the blood sugar was measured immediately. The fasting period lasted 24 hours or until signs of hypoglycemia as mentioned above or blood glucose below 3.0 mmol/L. Patients received an IV bolus of 10% glucose according to weight if signs of hypoglycemia occurred.

Analyses of blood samples and expired 13CO2. Venous blood was transferred to cooled tubes with EDTA (Ethylenediaminetetraacetic acid) (0.33M, 10μL mL-1) and spun at 4,000 rpm for 10 minutes. Plasma was distributed to Eppendorf tubes and immediately frozen on dry ice and stored at -80°C until analysis. Plasma insulin and glucagon analyses were performed at the Department of Clinical Biochemistry at Rigshospitalet, Copenhagen, Denmark (Cobas 8000, Roche, Rotkreuz Switzerland). Plasma free fatty acids and catecholamines were analyzed by spectrophotometry (Multiskan GO, Thermo Scientific, SkanIt™ Software, Thermo Fisher Scientific Inc., USA). Plasma palmitate, β-hydroxybuturate, acetoacetate, pyruvate, glycerol and amino acids as well as 13CO2-breath enrichment were analyzed by gas chromatography isotope ratio-mass spectrometry (Thermo Finnigan MAT GmbH, Bremen, Germany). Isotope tracer enrichments were determined using gas chromatography-mass spectrometry (Thermo Finnigan MAT GmbH, Bremen, Germany).

Glucose and lactate were analyzed on (ABL 700) immediately as the blood was drawn.

Shofield equation was used to calculate expected basal metabolic rate for the children: Males 10-17 years: (17.7 x weight+657+105) and females 10-17 years: (13,4 x weight+692+112) and the results were compared with the resting metabolic rate (RMR) measured by indirect calorimetric, as described above, at the end of the study, were patients had been resting and fasting for more than 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low skeletal muscle mass

Exclusion Criteria:

* Competing disorders interfering with interpretation of results
* Medication that will interfere with results
* Compliance problems
* Participation in other clinical trials that will interfere with interpretation of results
* Pregnancy or breastfeeding

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in fat metabolisms from fed to fasted state | 24 hours
  Using indirect calorimetri and stable isotope technique: of [U-13C]-palmitate (0.0026 mg kg-1 min-1, primed by a 0.085 mg kg-1 NaH13CO3 bolus) fat metabolism was measured at fed state and during 24 hours of fasting
Change in carbohydrates metabolisms from fed to fasted state | 24 hours
  Using indirect calorimetri and stable isotope technique: of [D2]-glucose (0.0728 mg kg-1 min-1, primed by a 3.203 mg kg-1 D2- glucose bolus) glucose metabolism was measured at fed state and during 24 hours of fasting

SECONDARY OUTCOMES:
Change in insulin, glucagon, epinephrine and norepinephrine and the metabolites palmitate, free fatty acids (FFA), glycerol, glucose, pyruvate, β-hydroxybuturate, acetoacetate from fed to fasted state. | 24 hours
  Hormones and metabolites were measured at fed state and during 24 hours of fasting
Change in glucagon from fed to fasted state. | 24 hours
  Glucagon was measured at fed state and during 24 hours of fasting
Change in epinephrine from fed to fasted state. | 24 hours
  Epinephrine was measured at fed state and during 24 hours of fasting
Change in norepinephrine from fed to fasted state. | 24 hours
  Norepinephrine was measured at fed state and during 24 hours of fasting
Change in palmitate from fed to fasted state. | 24 hours
  Palmitate was measured at fed state and during 24 hours of fasting
Change in free fatty acids (FFA) from fed to fasted state. | 24 hours
  FFA was measured at fed state and during 24 hours of fasting
Change in glycerol from fed to fasted state. | 24 hours
  Glycerol was measured at fed state and during 24 hours of fasting
Change in glucose from fed to fasted state. | 24 hours
  Glucose was measured at fed state and during 24 hours of fasting
Change in pyruvate from fed to fasted state. | 24 hours
  Pyruvate was measured at fed state and during 24 hours of fasting
Change in β-hydroxybuturate from fed to fasted state. | 24 hours
  β-hydroxybuturatewas measured at fed state and during 24 hours of fasting
Change in acetoacetate from fed to fasted state. | 24 hours
  Acetoacetate was measured at fed state and during 24 hours of fasting

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No